CLINICAL TRIAL: NCT00787566
Title: A Randomized, Single Administration, Double-blind, Parallel-group Phase 2 Dose Finding Study to Assess the Efficacy, Tolerability, and Safety of TRG (Intranasal Granisetron) in Patients With Chemotherapy-induced Nausea and Vomiting (CINV) Associated With the Administration of Highly Emetogenic Chemotherapy
Brief Title: Phase 2 Study of Efficacy, Tolerability, and Safety of Intranasal Granisetron for Chemo-Induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Nippon Biomedical Laboratories, Ltd. (Industry)
Responsible Party: Vanaja Ragavan, MD, Aviana Consulting, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TRG-002
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
Keywords: Highly emetogenic chemotherapy induced nausea and vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 0.5 mg of TRG (intranasal granisetron) (Experimental): 0.5 mg dose, intranasal powder, single spray, administered once
  Interventions: Drug: Intranasal granisetron
- 1.0 mg of TRG (intranasal granisetron) (Experimental): 1.0 mg dose, intranasal powder, songle spray, administered once
  Interventions: Drug: Intranasal granisetron
- 2.0 mg of TRG (intranasal granisetron) (Experimental): 2.0 mg dose, intranasal powder, single spray, administered once
  Interventions: Drug: Intranasal granisetron

INTERVENTIONS:
Drug: Intranasal granisetron — 0.5 mg, 1.0 mg or 2.0 mg dose of TRG prior to the administration of a highly-emetogenic chemotherapy regimen
  Other Names: TRG

SUMMARY:
Brief Summary: A randomized, single administration, double-blind, parallel- group Phase 2 dose finding study to assess the efficacy, tolerability, and safety of TRG in patients with chemotherapy-induced nausea and vomiting (CINV) associated with the administration of highly emetogenic chemotherapy.

Primary Objective: To select a dose for Phase 3 by assessing the efficacy, safety, and tolerability of 3 doses of TRG in patients with CINV associated with the administration of highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically and/or cytologically confirmed cancer
* ECOG performance status of 0, 1, or 2
* Patients with life expectancy of at least 3 months
* Patients who are chemotherapy naïve
* Patients who will be receiving the first cycle of a highly emetogenic regimen according to the MASCC criteria or the Hesketh criteria
* Patients with adequate metabolic or hematologic values for chemotherapy
* Patients with intact nasal mucosa
* Non child-bearing potential patients
* Patients able to read and write at a competent level, and capable of giving legal consent
* Patients who have provided written informed consent

Exclusion Criteria:

* Patients who do not receive a chemotherapy regimen which is a highly emetogenic chemotherapy regimen according to the MASCC or the Hesketh criteria
* Patients with nasal cancers, pharyngeal cancers, maxillary sinus cancers, or ethmoid sinus cancers
* Patients with nasal ulcers, septal perforation, or other nasal conditions that may interfere with IN administration
* Patients with any episode of retching, vomiting, or uncontrolled nausea within 48 hours before dosing with TRG and/or administration of chemotherapy
* Patients who have received radiation therapy in the 14 days before dosing with TRG, or for whom radiation therapy is scheduled during the 7 days after a TRG dose
* Patients who have received any investigational product within 30 days prior to study entry
* Patients who have received any drug or who were scheduled to receive any drug with antiemetic efficacy within 24 hours of the start of treatment
* Patients who have an allergy or hypersensitivity to granisetron or other selective 5hydroxytryptamine3(5-HT3) receptor antagonists
* Patients with ECOG performance status of 3 or 4
* Patients who have or have a history of brain tumors, head cancers, or neck cancers
* Patients who have a psychological problem that, in the Investigator's opinion, is severe enough to interfere with study eligibility or with interpretation of study results
* Patients who are pregnant (urine test) or breastfeeding
* Patients who have received prior cytotoxic chemotherapy given for the treatment of cancer
* Patients scheduled to receive multiple day chemotherapy
* Patients with clinically relevant abnormal laboratory values at the discretion of the Investigator
* Patients with clinically relevant hepatic, renal, infectious, neurological, or psychiatric disorders, or any other major systemic illness at the discretion of the Investigator
* Patients with any prevalence or cause of nausea and vomiting other than chemotherapy
* Patients using systemic steroids for any indication, or patients using steroids other than dexamethasone for prevention of chemotherapy-induced nausea and vomiting, or patients using dexamethasone for chemotherapy-induced nausea and vomiting at doses other than recommended in the MASCC antiemetic guidelines
* Patients with a QT interval greater than 500 ms or with acute ischemic changes or cardiac abnormality predisposing to arrhythmia on screening electrocardiogram (ECG) or by history
* Patients with a history of drug and/or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The study is conducted at 14 Centers, in 14 cities accross the United States, The Study Is Managed by Kendle International, in Wilmington, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.0 mg of TRG (Intranasal Granisetron): 1.0 mg dose, intranasal powder, single spray, administered once
Period: Overall Study
Arm/Group | 0.5 mg of TRG (Intranasal Granisetron) | 1.0 mg of TRG (Intranasal Granisetron) | 2.0 mg of TRG (Intranasal Granisetron)
Started | 21 | 25 | 22
Completed | 21 | 24 (1 patient withdrew from the study due to an AE related to chemotherapy agent administration.) | 22
Not Completed | 0 | 1 | 0
Not completed — AE related to chemotherapy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg of TRG (Intranasal Granisetron) | 1.0 mg of TRG (Intranasal Granisetron) | 2.0 mg of TRG (Intranasal Granisetron) | Total
Number analyzed (Participants) | 21 | 25 | 22 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 14 | 45
  >=65 years | 7 | 8 | 8 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (15.9) | 60.0 (10.2) | 61.0 (12.0) | 58.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 17 | 53
  Male | 2 | 8 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 21 | 25 | 22 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Control
Description: Complete Control is defined as no emetic episodes, no use of rescue medications, and no more than mild nausea as defined by a categorial scale.
Time Frame: 24 hours
Population: ITT population
Measure: Number; unit: Percentage
Arm/Group | 0.5 mg of TRG (Intranasal Granisetron) | 1.0 mg of TRG (Intranasal Granisetron) | 2.0 mg of TRG (Intranasal Granisetron)
Number analyzed (Participants) | 21 | 25 | 22
Percentage | 71.4 | 76.0 | 90.9

2. Secondary Outcome: Percentage of Patients With Complete Response
Description: Complete Response is defined as no emetic episodes and no use of rescue medications
Time Frame: 24 hours
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Patients With Total Response
Description: Total Response is defined as no nausea, no emetic episodes, and no use of rescue medications
Time Frame: 24 hours
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Patients With Major Control of Emesis
Description: Major Control of emesis = 2 emetic episodes
Time Frame: 24 hrs
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Patients With Minor Control of Emesis
Description: Minor Control of emesis: 3-5 emetic episodes
Time Frame: 24 hrs
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Patients With Failure
Description: Failure: > 5 emetic episodes
Time Frame: 24 hrs
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Patients Using Rescue Medications
Time Frame: 24 hours
Reporting Status: Not Posted

8. Secondary Outcome: Time to First Emetic Episode
Time Frame: 24 hours
Reporting Status: Not Posted

9. Secondary Outcome: Time to First Rescue Medication
Time Frame: 24 hours
Reporting Status: Not Posted

10. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is based on time to first emetic episode or time to rescue medication, whichever occurs first
Time Frame: 24 hours
Reporting Status: Not Posted

11. Secondary Outcome: Number of Emetic Episodes
Time Frame: 24 hours
Reporting Status: Not Posted

12. Secondary Outcome: Severity of Nausea Measured by a 4 Categorical Scale
Description: 4 categorical scale: none, mild (did not interfere with normal daily life), moderate (interfered with normal daily life), and severe (bedridden due to nausea/ required the patient to be bedridden)
Time Frame: 24 hours
Reporting Status: Not Posted

13. Secondary Outcome: Patient Global Satisfaction With Antiemetic Therapy Measured by a VAS
Description: VAS (visual analog scale) 0: not at all satisfied, 100: totally satisfied
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Dosing of study drug through safety follow-up period (maximum 38 days)
Description: Telephone questioning 2-24 hours after start of chemotherapy; 8 day patient diary
Arm/Group | 0.5 mg of TRG (Intranasal Granisetron) | 1.0 mg of TRG (Intranasal Granisetron) | 2.0 mg of TRG (Intranasal Granisetron)
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/25 | 1/22
Other Adverse Events (participants affected / at risk) | 16/21 | 16/25 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg of TRG (Intranasal Granisetron) (N=21) | 1.0 mg of TRG (Intranasal Granisetron) (N=25) | 2.0 mg of TRG (Intranasal Granisetron) (N=22)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to study mediation
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to study medication
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Not related to study medication
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to study medication
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to study medication
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to study medication
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to study medication
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg of TRG (Intranasal Granisetron) (N=21) | 1.0 mg of TRG (Intranasal Granisetron) (N=25) | 2.0 mg of TRG (Intranasal Granisetron) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Fatigue (General disorders) | 8 (8) | 6 (6) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Weight decrease (Investigations) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SNBL and investigators agreed that SNBL would retain the exclusive right to disseminate data arising from the study through either publication or presentation, including study results, and that SNBL would retain exclusive editorial rights over manuscripts or presentations.